CLINICAL TRIAL: NCT07363044
Title: A Prospective Randomised Study of Treatment Selection Based on Epigenetic Markers Versus Standard of Care Treatment Selection in Adults With CROHN's Disease
Acronym: OMICROHN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alimentiv Inc. (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Horizon Europe (Unknown); Stichting Amsterdam UMC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT-01727
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease (CD)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigator-Guided Treatment Arm (Other)
  Interventions: Other: Investigator-Guided Treatment Arm
- Epigenome-Guided Treatment Arm (Experimental)
  Interventions: Device: Epigenome-Guided Treatment Arm

INTERVENTIONS:
Device: Epigenome-Guided Treatment Arm — Participants will receive UST or VDZ biologic therapy as indicated by an epigenome read-out of peripheral blood using a hybrid capture-based methylation assay. The assay and EpiPredict software will indicate the probability of response to VDZ and UST. The biologic with the predicted highest likelihood of success will be communicated to the investigator and the biologic initiated using standard dosing regimens.
  Arms: Epigenome-Guided Treatment Arm
Other: Investigator-Guided Treatment Arm — Assigned to UST or VDZ per conventional SOC and without the use or knowledge of epigenome results.
  Arms: Investigator-Guided Treatment Arm

SUMMARY:
This is a multicentre, prospective, randomised, controlled, open-label study to assess the efficacy, safety, and cost-effectiveness of epigenome-guided treatment selection compared to usual standard-of-care (SOC) treatment selection in patients initiating biologic therapy for the treatment of their active Crohn's Disease (CD).

DETAILED DESCRIPTION:
This trial will include 378 participants with active CD, defined as an HBI > 6 and the presence of endoscopic ulceration. Approximately 50% of the enrolled population will be bio-naïve and 50% exposed to no more than 1 prior biologic.

Eligible participants will be randomised 1:1 to either epigenome-guided treatment selection or usual SOC treatment selection. Randomization will be stratified by prior biologic use (yes/no) and corticosteroid use (yes/no) at baseline.

Blood samples for the assessment will be collected for all participants during screening. Peripheral blood will be tested via a machine-learning-powered epigenetic biomarker assay. EpiPredict is a software designed for CSV file input, data transfer, storage, and display, and will be serving as a EpiPredict clinical decision support system. It recommends treatment selections for 2 biologics (Vedolizumab (VDZ) and Vedolizumab (UST)) for CD utilizing genetic data.

The intervention (EpiPredict software) will indicate the probability of response to both VDZ and UST (though sites will only be provided with the treatment with the highest outcome) for the treatment of CD using a hybrid capture-based methylation assay (approved for research use only) and the EpiPredict software.

All participants in the study will be administered their biologic therapy in accordance with the product label and local SOC recommendations. Dose adjustments will be allowed in both groups at the treating investigator's discretion.

During the 26-week treatment period, the study assessments will follow the SOC regimen of the assigned biologic treatment. For participants receiving VDZ, study assessments are to occur at Weeks 6, 14, and 26; for participants receiving UST, study assessments are to occur at Weeks 8, 16, and 26.

Long-term follow up assessments are to occur every 6 months (Months 12, 18, and 24) after Week 26. Data for long-term follow up assessments will be collected from the participant's medical records captured at routine SOC visits and online questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria for enrolment into the study:

1. Aged 18 years or older at the time of informed consent.
2. Documented diagnosis of ileal, ileocolonic, or colonic CD (may be confirmed at baseline study endoscopy).
3. Active CD, as defined by HBI > 6 and SES-CD ≥ 6 for colitis/ileocolitis and ≥ 4 for ileitis only.
4. Eligible to receive either VDZ and/or UST therapy for the treatment of CD per the approved drug label requirements and in the opinion of the treating physician.
5. Must meet all eligibility criteria for biologic therapy initiation as per local SOC, including absence of chronic/opportunistic infections as demonstrated by local protocols for human immunodeficiency virus, tuberculosis, active cytomegalovirus, hepatitis B and C, and Clostridioides difficile infection. Local vaccination protocols apply as per SOC.
6. Nonpregnant and nonlactating. Participants of childbearing potential must agree to follow local SOC guidelines for use of biologics in pregnancy/lactation, including appropriate contraception, during the study; must agree to avoid becoming pregnant from the time of informed consent up until Week 26.
7. If receiving nonbiologic therapies for inflammatory bowel disease, including thiopurines and methotrexate, must have initiated at least 3 months prior to screening and must be on a stable dose for at least 2 weeks prior to screening.
8. If receiving oral corticosteroids, the participant is eligible if they meet all the following criteria:

   * The dose is up to a maximum of prednisone ≤ 40 mg/day or budesonide ≤ 9 mg/day or equivalent.
   * The dose has been stable for ≥ 2 weeks prior to screening.
   * The participant is willing to initiate a corticosteroid taper within 2 weeks after initiating biologic treatment.
9. In the opinion of the investigator, the participant is able to understand and comply with protocol requirements including treatment as assigned per the protocol.
10. Able to participate fully in all aspects of this clinical study. Full comprehension of consent language and informed consent must be obtained from the participant, or the participant's legally acceptable representative, and documented

Exclusion Criteria:

Participants who meet any of the following criteria are to be excluded from the study:

1. Prior treatment with VDZ or UST.
2. Prior treatment with more than 1 advanced therapy (eg, any biologic [ie, anti- tumour necrosis factor (TNF), anti-interleukin, anti-integrin]) or advanced oral small molecule [ie, Janus kinase inhibitor]) for CD.
3. CD-related complications that in the opinion of the investigator would interfere with participation in the study, including but not limited to:

   * Ileorectal anastomosis (rectum < 15 cm), or a proctocolectomy.
   * Short bowel syndrome.
   * All ostomies.
   * Symptomatic strictures in the bowel or symptomatic strictures in the ileum or ileocecal valve that have a stenosis.
   * Suspected or diagnosed active intra-abdominal or perianal abscess that have not been appropriately treated.
4. History or current diagnosis of ulcerative colitis (unless this diagnosis was made erroneously), indeterminate colitis, idiopathic colitis (ie, colitis not consistent with CD), microscopic colitis, or colonic mucosal dysplasia (excluding dysplasia in resected adenomas).
5. Increased risk of infectious complications (eg, recent pyogenic infection, any congenital or acquired immunodeficiency, or past organ, bone marrow, or stem cell transplantation).
6. Any topical rectal therapy for treatment of CD within 2 weeks prior to the screening endoscopy.
7. Nonsteroidal anti-inflammatory drugs (NSAIDs) as chronic treatment, except for cyclooxygenase-2logic selective NSAIDS (celecoxib).
8. Faecal microbiota transplant (includes human microbiota-based therapeutics) within 4 weeks prior to randomisation.
9. Any major surgery (in the investigator's opinion) performed within 8 weeks prior to randomisation or planned during the study.
10. History of excessive alcohol or drug abuse that, in the opinion of the investigator, may interfere with the participant's ability to comply with the study procedures.
11. Serious underlying disease other than CD that in the opinion of the investigator may interfere with the participant's ability to participate fully in the study or would compromise participant safety (such as history of malignancies, major neurological disorders, any unstable or uncontrolled medical disorder, or any known or suspected contraindication to any of the study biologics according to local prescribing information).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of epigenome-guided treatment selection to usual SOC treatment selection for inducing clinical remission and endoscopic response at Week 26 in participants with active CD. | Baseline to Week 26
  Corticosteroid-free clinical remission (Harvey-Bradshaw Index [HBI] score ≤ 4) and endoscopic response (≥ 50% decrease from baseline in the Simple Endoscopic Score for Crohn's Disease [SES-CD])

SECONDARY OUTCOMES:
To explore the optimal threshold of EpiPredict results in predicting treatment response using data from participants assigned to the epigenome-guided treatment selection group | Baseline to Week 26
  Receiver-operating characteristic curve area analysis will be used Predicted likelihood of success of reaching corticosteroid-free clinical remission and endoscopic response
To compare the efficacy of epigenome-guided treatment selection to usual SOC treatment selection for improving clinical and endoscopic outcome measures at Week 26 in participants with active CD | Baseline to Week 26
  Endoscopic response (≥ 50% decrease from baseline in SES-CD score) Endoscopic remission (SES-CD ≤ 3) Clinical remission (HBI ≤ 4) Corticosteroid-free clinical remission Clinical response (decrease in HBI ≥ 3 points from baseline) Corticosteroid-free deep remission (HBI ≤ 4 and SES-CD ≤ 3)
To evaluate the cost-effectiveness of epigenome-guided treatment selection compared to usual SOC treatment selection | Baseline to 24 Months
  Societal costs as measured by the modified iMTA Medical Cost Questionnaire and modified iMTA Productivity Cost Questionnaire questionnaires Quality of life-years as measured by the European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) questionnaire

OTHER OUTCOMES:
To assess the safety of a treatment based on epigenome-guided treatment selection compared to usual SOC treatment selection | Baseline to Week 26
  Adverse events CD-related complications, hospitalisations, and/or surgeries
To explore additional efficacy measures of epigenome-guided treatment selection compared to usual SOC treatment selection at Week 26 in participants with active CD. | Baseline to Week 26
  Achieving a minimally clinically important difference in patient-reported health-related quality of life (HRQOL) compared to baseline as measured by the EQ-5D-5L Clinical remission (HBI ≤ 4) Clinical response (decrease in HBI ≥ 3 points from baseline) Clinical remission (Crohn's Disease Activity Index [CDAI] score of < 150) over time Time to symptomatic remission (HBI ≤ 4) No drainage on gentle finger compression in participants with draining fistulas Extra-intestinal manifestations Histologic response, as defined in the statistical analysis plan (SAP) Histologic remission, as defined in the SAP Whether the participant achieved 25%, 50%, and 75% reduction from baseline in the Robarts Histopathology Index (RHI) score Serum trough concentrations of biologic drug Biochemical remission CRP ≤ 5.0 mg/L and/or fecal calprotectin [FC] < 250 µg/g) Change in the Symptoms and Impact Questionnaire-CD (SIQ-CD) score
In a subset (~30%) of participants, to evaluate response by intestinal ultrasound (IUS) in participants assigned to epigenome-guided treatment selection compared to usual SOC treatment selection | Baseline to Week 26
  Proportion of participants with IUS response (defined as by reduction in bowel wall thickness [BWT > 25%] or [> 2.0 mm] or [> 1.0 mm and one colour Doppler signal (CDS) reduction]) Proportion of participants with transmural remission (defined by BWT ≤ 3 mm and normal/0 CDS) Proportion of participants with transmural remission and endoscopic remission

CONTACTS AND LOCATIONS:
Locations (30):
- Belgium (13):
  - Imeldahospital, Bonheiden
  - AZ Klina, Brasschaat
  - H.U.B. - Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem
  - AZ Maria Middelares, Ghent
  - AZ Sint Lucas, Ghent
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire (CHU) de Liege, Liège
  - Groupe sante CHC/Clique du MontLegia, Liège
  - AZ Oostende, Ostend
  - AZ Delta VZW, Roeselare
  - CHU UCL Namur asbl Site Godinne, Yvoir
- IRCCS Ospedale San Raffaele, Milan, Italy
- Netherlands (6):
  - Amsterdam UMC, Amsterdam
  - OLVG Oost, Amsterdam
  - Maastricht UMC, Maastricht
  - Radboudumc, Nijmegen
  - Elisabeth-TweeSteden Ziekenhuis (ETZ), Tilburg
  - Universitair Medisch Centrum Utrecht, Utrecht
- United Kingdom (10):
  - Northern Care Alliance - Fairfield General Hospital, Bury
  - Cambridge University Hospitals NHS Trust, Cambridge
  - Hull University Teaching Hospital NHS Trust, Cottingham
  - The Dudley Group NHS Foundation Trust, Dudley
  - Cardiff & Vale UHB, Llandough
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Hampshire Hospital NHS Foundation Trust, Winchester